CLINICAL TRIAL: NCT01409603
Title: A Phase I, Open-Label, Randomized 3-Period Crossover Study in Healthy Male Subjects to Evaluate the Pharmacodynamic Interactions Between YM150 on Naproxen at Steady-State
Brief Title: To Evaluate Whether Naproxen and Darexaban (YM150) Interact in Their Effects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: 150-CL-039; 2009-015762-64 (EudraCT Number)
Record Dates: First submitted 2011-08-01; First posted 2011-08-04 (Estimated); Last update posted 2013-04-11 (Estimated); Status verified 2013-04

CONDITIONS: Pharmacodynamic Interaction; Healthy Subjects
Keywords: Pharmacodynamics; darexaban; naproxen; YM150; Phase 1
MeSH Terms: interventions — darexaban; Naproxen

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (6):
- Treatment arm A (Experimental): darexaban, wash-out, naproxen, wash-out, combination therapy
  Interventions: Drug: darexaban; Drug: Naproxen
- Treatment arm B (Experimental): darexaban, wash-out, combination therapy, wash-out, naproxen
  Interventions: Drug: darexaban; Drug: Naproxen
- Treatment arm C (Experimental): naproxen, wash-out, darexaban, wash-out, combination therapy
  Interventions: Drug: darexaban; Drug: Naproxen
- Treatment arm D (Experimental): naproxen, wash-out, combination therapy, wash-out, darexaban
  Interventions: Drug: darexaban; Drug: Naproxen
- Treatment arm E (Experimental): combination therapy, wash-out, naproxen, wash-out, darexaban
  Interventions: Drug: darexaban; Drug: Naproxen
- Treatment arm F (Experimental): combination therapy, wash-out, darexaban, wash-out, naproxen
  Interventions: Drug: darexaban; Drug: Naproxen

INTERVENTIONS:
Drug: darexaban — oral
  Other Names: YM150
Drug: Naproxen — oral
  Other Names: Naprosyne

SUMMARY:
The primary objective of this study is to evaluate whether naproxen and darexaban which have different effects on blood coagulation influence each other in their effects. Also it will be investigated whether the blood levels of either drug are influenced by the presence of the other drug. In addition, the safety and tolerability of each drug and the combination of the drugs will be investigated.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) between 18.5-30.0 kg/m2
* Male subjects must be non-fertile, i.e. surgically sterilized or must practice an adequate contraceptive method to prevent pregnancies

Exclusion Criteria:

* Known or suspected hypersensitivity to darexaban or naproxen or any components of the formulation used
* A contra-indication for the use of naproxen
* Any of the liver function tests (i.e. ALT, AST and bilirubin) above the upper limit of normal at repeated measures
* Any clinically significant history of any other disease or disorder - gastrointestinal, cardiovascular, respiratory, renal, hepatic, neurological, dermatological, psychiatric or metabolic as judged by the medical investigator.
* Any clinically significant abnormality following the investigator's review of the pre-study physical examination, ECG and clinical laboratory tests
* Use of any prescribed or OTC (over-the-counter) drugs (including vitamins, natural and herbal remedies, e.g. St. John's wort) in the 2 weeks prior to admission to the Clinical Unit, except for occasional use of paracetamol (up to 3 g/day)
* Regular use of any inducer of liver metabolism (e.g. barbiturates, rifampicin) in the 3 months prior to admission to the Clinical Unit
* Donation of blood or blood products within 3 months prior to admission to the Clinical Unit
* Any use of drugs of abuse, or smoking of more than 10 cigarettes (or equivalent) or more than 21 units (210 g) of alcohol per week within the 3 months prior to study
* Participation in any clinical study within 3 months or participation in more than 3 clinical studies within 12 months, prior to the expected date of enrolment into the study, provided that the clinical study did not entail a biological compound with a long terminal half life

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2010-01; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

PRIMARY OUTCOMES:
Assessment of pharmacodynamics of naproxen | Baseline and 3 hours after multiple dosing (darexaban: 6 days, naproxen: 4 days) of darexaban, naproxen, or a combination of the two

SECONDARY OUTCOMES:
Assessment of pharmacodynamics of darexaban | Baseline and 3 hours after multiple dosing (darexaban: 6 days, naproxen: 4 days) of darexaban, naproxen, or a combination of the two
Pharmacokinetics of darexaban assessed by plasma concentration | Plasma samples are taken until 24 hours after six days of dosing of darexaban, or the combination with naproxen
Pharmacokinetics of naproxen assessed by plasma concentration | Plasma samples are taken until 12 hours after four days of dosing of naproxen, or the combination with darexaban
Monitoring of safety and tolerability through assessment of vital signs, Electrocardiogram (ECG), clinical safety laboratory and adverse events | 6 days (for treatment periods with darexaban) or 4 days. (naproxen alone)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Study Manager, Study Chair — Astellas Pharma Europe B.V.; Principal Investigator, Principal Investigator — SGS Aster, Paris, France
Locations (1):
- SGS Aster, Paris, France